CLINICAL TRIAL: NCT07380516
Title: Adoption of the Xo-Motion R in the Subacute and Chronic SCI Populations at the Glenrose Rehabilitation Hospital
Brief Title: Xo-Motion R Exoskeleton in SCI-Adoption Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Praxis Spinal Cord Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00159509
Record Dates: First submitted 2025-12-02; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Spinal Cord Injury
Keywords: exoskeleton; rehabilitation; locomotion; SCI
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inpatient SCI Group (Other): During their inpatient rehabilitation, the XoMotionR will be incorporated into their locomotor therapy program for approximately 30-45minutes, 2-3 times per week, up to 6 weeks. Inpatient intervention will be focused on promoting early weight-bearing, postural control, and initiation of step cycles. Training includes progressive walking tasks that emphasize symmetrical lower limb loading, upright posture, and engagement of trunk musculature. In addition to forward ambulation, sessions incorporate functional activities such as sit-to-stand transitions, pivot turns, and standing balance tasks which are all possible with the self-balancing XoMotion-R. The intervention is individualized based on tolerance, cardiovascular response, and patient progress, with adjustments made to walking speed, step length, and assistance levels over time.
  Interventions: Device: XoMotionR- assisted locomotor training
- Outpatient SCI Group (Other): Through our Specialized Outpatient Rehabilitation Program or Research Lab in the Courage Centre, SCI outpatients will be recruited and the XoMotionR will be incorporated into their locomotor therapy program for approximately 30-45minutes, 2-3 times per week, up to 6 weeks. Outpatient intervention will follow a task-specific approach emphasizing increased walking distance, reduced exoskeleton assistance, and advancement toward community-based ambulation goals. In this phase, the focus shifts toward higher-level gait tasks, including multi-surface walking, obstacle negotiation, and endurance training. Individuals are encouraged to use assistive devices with progressively less support as their neuromuscular control improves.
  Interventions: Device: XoMotionR- assisted locomotor training

INTERVENTIONS:
Device: XoMotionR- assisted locomotor training — The XoMotion-R self-balancing exoskeleton will be utilized for locomotor training in both the inpatient and outpatient setting. Inpatient intervention will be focused on promoting early weight-bearing, postural control, and initiation of step cycles. Training includes progressive walking tasks that emphasize symmetrical lower limb loading, upright posture, and engagement of trunk musculature. In addition to forward ambulation, sessions incorporate functional activities such as sit-to-stand transitions, pivot turns, and standing balance tasks which are all possible with the self-balancing XoMotion-R. The intervention is individualized based on tolerance, cardiovascular response, and patient progress, with adjustments made to walking speed, step length, and assistance levels over time.
  Outpatient intervention will follow a task-specific approach emphasizing increased walking distance, reduced exoskeleton assistance, and advancement toward community-based ambulation goals. In this phase,

SUMMARY:
After spinal cord injury (SCI), many people lose their ability to walk and do not have access to equipment and assistance that could help them regain functional abilities. Furthermore, many who have the potential to regain function are further hindered by a loss of function in their upper body that limits their ability to use a walker or crutches, thus eliminating options for mobility.

This study seeks to determine the safety and feasibility of the XoMotion-R, a self-balancing exoskeleton that allows people with American Spinal Injury Association Impairment Scale (AIS) rating of B-D SCI to walk hands-free in inpatient and outpatient settings. This study will examine how use of the XoMotion-R affects functional outcomes and identify setting-specific barriers and facilitators to clinical adoption.

This single-arm feasibility study will recruit 8 SCI inpatients and 8 SCI outpatients whose goal is to improve their walking and incorporate the XoMotion-R into their rehabilitation sessions. Participants will work on a variety of gait tasks tailored to their functional level. The goal is to determine whether early robotic gait training can improve functional outcomes and decrease length of stay, secondary complications, and long-term disability burden.

ELIGIBILITY:
Inclusion Criteria:

* SCI (AIS C or D in inpatient setting, AIS B-D in outpatient setting; inclusive of cervical injuries)
* inpatients who are preambulatory with predicted probability of walking independently 1year after injury >50% (Hicks et al., 2017)
* outpatients with a functional goal of improved locomotion where the XoMotion is clinically suited to support the achievement of their functional goals

Exclusion Criteria:

* SCI AIS A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
SCI Standing and Walking Assessment (SWAT) | Baseline and completion of 6 weeks of locomotor therapy with the XoMotionR
  The SWAT will be the primary effectiveness outcome for the inpatient group.
6min Walk Test (6MT) (Outpatient group) | Baseline and completion of 6 weeks of locomotor therapy with the XoMotionR
10-m Walk Test (10MWT) (Outpatient Group) | Baseline and completion of 6 weeks of locomotor therapy with the XoMotionR
Modified Timed Up and Go (mTUG) (Outpatient Group) | Baseline and completion of 6 weeks of locomotor therapy with the XoMotionR
Berg Balance Scale (BBS) (Outpatient Group) | Baseline and completion of 6 weeks of locomotor therapy with the XoMotionR

SECONDARY OUTCOMES:
Device-generated metrics (Number of steps taken) | Throughout study completion, for an average of 6 weeks
Device-generated metrics (Level of assistance provided) | Throughout study completion, for an average of 6 weeks

OTHER OUTCOMES:
Functional Independence Measure (FIM) | Baseline and completion of 6 weeks of locomotor therapy with the XoMotionR
SCIM III | Baseline and completion of 6 weeks of locomotor therapy with the XoMotionR
System Usability Scale (SUS) | At 6 weeks
  The SUS is a standard scale used to evaluate a technology. It will be completed by all clinicians who used the device at the end of the study.
Participant Structured Interview | At 6 weeks
  Structured interview to accurately capture the participants overall experience and impressions with the exoskeleton.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica M D'Amico, PhD, Principal Investigator — University of Alberta and Alberta Health Services
Locations (1):
- Glenrose Rehabilitation Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No